CLINICAL TRIAL: NCT01861184
Title: A Study of Pneumococcal Carriage in Hospitalised Patients With Lower Respiratory Tract Infections
Brief Title: Pneumococcal Carriage in Patients With Lower Respiratory Tract Infection (LRTI)
Status: Completed | Type: Observational
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 100090090
Record Dates: First submitted 2013-05-21; First posted 2013-05-23 (Estimated); Last update posted 2022-06-09 (Actual); Status verified 2013-05

CONDITIONS: Lower Respiratory Tract Infections
Keywords: Lower respiratory tract infection; LRTI; Pneumococcal carriage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples Nasal wash samples Nasopharyngeal swabs (where nasal wash not possible) Urine samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LRTI group: Non-pneumonic LRTI (no radiological consolidation but the presence of clinical signs) or community acquired pneumonia (radiological consolidation) Able to give fully informed consent (mental capacity assessed using trust guidelines) Age>18yrs old Fluent English speaker
- Control group: Able to give fully informed consent (mental capacity assessed using trust guidelines) Age>18yrs old Fluent English speaker

SUMMARY:
We are interested in developing new and better ways of diagnosing the cause of lower respiratory tract infections including pneumonia. Currently we find the causal bug (bacteria or virus) in less than 50% of patients with pneumonia. A potential way to better find the bug responsible may include checking for bugs in the nose by a nasal wash or swab. Better diagnostics would allow more targeted antibiotic therapy and in the future this technique may be used as a way of checking the efficiency of new vaccines.

We are recruiting both patients with respiratory infections and also a 'control' group of patients admitted to hospital who do not have respiratory infection. We need to have access to your medical history information to make sure you are eligible and suitable for the study. If you participate in the study, it is important that the study doctors continue to have access to your personal Investigator Designation Contact telephone Dr Andrea Collins PhD student/research SpR xxxxxxxxxxxxx Carole Hancock Research nurse 0151 706 4856 Prof Stephen Gordon Principle Investigator 0151 705 3169 NW PIL V1.3: October 2012 REC ref: 12/NW/0713 information so you can be followed up properly and so we can contact you during the study if needed.

Patients in both groups will have a nasal wash (or swab), blood (30mls = 6 teaspoons) and urine taken on the day of recruitment and a nasal wash (or swab) and blood (30mls = 6 teaspoons) taken 6 weeks later (this is likely to be as an out-patient at the Royal Liverpool, in extreme circumstances this will occur at the patient's home).

DETAILED DESCRIPTION:
STUDY DESIGN OVERVIEW

Overall research aim

To analyse pneumococcal carriage rates in patients hospitalised with LRTI.

Primary endpoint

Rate of pneumococcal carriage in patients hospitalised with LRTI and age matched controls.

Secondary endpoints

1. Density of pneumococcal carriage in patients hospitalised with LRTI and age matched controls
2. Alterations of T cell function (Th1, Th17, T regs) in LRTI patients and age matched controls (versus younger adults as part of our existing 'P4' study).

Study design Patients hospitalised with LRTI between November 2012 and April 2014 will be approached within 72 hours of admission.

Patients recruited into the study will consist of those hospitalised with LRTI and a control group of age matched patients (within +/- 10 years) hospitalised for reasons other than respiratory infection.

ELIGIBILITY:
Inclusion criteria for LRTI patients:

Non-pneumonic LRTI (no radiological consolidation but the presence of clinical signs) or community acquired pneumonia (radiological consolidation) Able to give fully informed consent (mental capacity assessed using trust guidelines) Age>18yrs old Fluent English speaker

Exclusion criteria for LRTI patients:

Infective exacerbation of COPD or bronchiectasis without consolidation Oxygen saturations <86% on air Tuberculosis suspected Neutropenia

Inclusion criteria for controls:

Able to give fully informed consent (mental capacity assessed using trust guidelines) Age>18yrs old

* 10 years of recruited LRTI patient Fluent English speaker

Exclusion criteria for controls:

Signs/symptoms of respiratory infection Oxygen saturations <86% on air Neutropenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the hospital with Lower Respiratory Tract Infection
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Rate of pneumococcal carriage in patients hospitalised with LRTI and age matched controls. | 6weeks
  Pneumococcal colonisation will be defined based on the culture (+/-PCR) result of nasal wash/NPS taken at day 0 and 6 weeks.

SECONDARY OUTCOMES:
Density of pneumococcal carriage in patients hospitalised with LRTI and age matched controls | 6weeks
  Density will be determined using a modified version of Miles and Misra dilutions.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Stephen Gordon, Principal Investigator — Royal Liverpool University Hospital/ Liverpool School of Tropical Medicine
Locations (1):
- Royal Liverpool University Hospital, Liverpool, United Kingdom

REFERENCES:
- [Derived] German EL, Al-Hakim B, Mitsi E, Pennington SH, Gritzfeld JF, Hyder-Wright AD, Banyard A, Gordon SB, Collins AM, Ferreira DM. Anti-protein immunoglobulin M responses to pneumococcus are not associated with aging. Pneumonia (Nathan). 2018 Jun 5;10:5. doi: 10.1186/s41479-018-0048-3. eCollection 2018. PMID 29992080